CLINICAL TRIAL: NCT05797155
Title: A Mobile App Based Cognitive Dissonance Intervention for Smoking Cessation
Acronym: Support2Quit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Behavioral Intervention Strategies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DP006495-02
Record Dates: First submitted 2023-03-09; First posted 2023-04-04 (Actual); Results first posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Intervention Model Description: This study will recruit 500 daily adult smokers through social media to test the Support2Quit app for smoking cessation. Participants will be randomly assigned to either the Support2Quit app or an app that has similar content but no tasks for inducing cognitive dissonance among participants.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Support2Quit App - Cognitive Dissonance Based Smoking Cessation (Experimental): This group will receive daily smoking cessation tips and will be asked to complete activities within the app that are designed to induce cognitive dissonance, create and share videos related to the activities with an online group, and provide support to other group members
  Interventions: Behavioral: Support2Quit App - Cognitive Dissonance Based Smoking Cessation + Smoking Cessation Tips
- Comparison App - Smoking Cessation Support without Cognitive Dissonance Activities (Active Comparator): This group will use an app that consists of tips for quitting cigarettes but does not include the cognitive dissonance component.
  Interventions: Behavioral: Tips for Smoking Cessation App

INTERVENTIONS:
Behavioral: Support2Quit App - Cognitive Dissonance Based Smoking Cessation + Smoking Cessation Tips — Support2Quit App (Cognitive Dissonance Based Smoking Cessation) Use of the Support2Quit app, completion of cognitive dissonance activities, sharing of videos with online group, and providing support to other group members
  Arms: Support2Quit App - Cognitive Dissonance Based Smoking Cessation
Behavioral: Tips for Smoking Cessation App — App containing daily tips for smoking cessation
  Arms: Comparison App - Smoking Cessation Support without Cognitive Dissonance Activities

SUMMARY:
This research study aims to develop a cognitive dissonance-based mobile app for smoking cessation (Support2Quit) and test the efficacy of the app with 500 adult smokers who express a desire to quit smoking.

DETAILED DESCRIPTION:
This research project will evaluate the Support2Quit mobile app for smoking cessation by having 500 daily adult smokers recruited through social media and randomized to either the Support2Quit app or an app that has similar content but no tasks for inducing cognitive dissonance among participants. Outcomes will be measured at 1- and 3-months post-baseline and will include quit attempts, number of days without smoking (smoke free days), and changes in smoking attitudes and behavior, and smoking abstinence. Usability data, system log data on program use, and participant satisfaction data will also be analyzed.

The researchers hypothesize that individuals using the cognitive dissonance intervention (CDI) will show greater increases in quit attempts, smoke free days, quit rates, and positive smoking attitudes and behaviors than individuals in the active comparison condition. The researchers will test whether gender, smoking dependence, readiness to quit, previous quit attempts, age of smoking initiation, and socio-economic status moderate intervention effects on smoking outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Self-reported daily smoking
* Having a valid home mailing address in the United States
* English-speaking
* Access to a smart phone with video capability for the duration of the project
* Expressed desire to quit smoking

Exclusion criteria:

• Currently participating in a tobacco cessation program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana Smith, PhD, Principal Investigator — Oregon Research Behavioral Intervention Strategies, Inc.
Locations (1):
- Oregon Research Behavioral Intervention Strategies, Inc., Springfield, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Support2Quit App - Cognitive Dissonance Based Smoking Cessation | Comparison App - Smoking Cessation Support without Cognitive Dissonance Activities
Started | 292 | 145
Completed | 259 | 133
Not Completed | 33 | 12
Not completed — Lost to Follow-up | 33 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Support2Quit App - Cognitive Dissonance Based Smoking Cessation | Comparison App - Smoking Cessation Support Without Cognitive Dissonance Activities | Total
Number analyzed (Participants) | 292 | 145 | 437
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.21 (12.00) | 48.84 (11.50) | 49.08 (11.82)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 215 | 104 | 319
  Male | 76 | 38 | 114
  Transgender | 1 | 1 | 2
  Non-binary | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 12 | 29
  Not Hispanic or Latino | 275 | 133 | 408
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 3 | 9
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 32 | 13 | 45
  White | 224 | 119 | 343
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 24 | 9 | 33
Region of Enrollment [Number; unit: participants]
  United States | 292 | 145 | 437
Highest level of education [Count of Participants; unit: Participants]
  Did not graduate high school | 12 | 1 | 13
  High school graduate | 63 | 23 | 86
  Some college, no degree | 91 | 44 | 135
  Technical school or associate degree | 52 | 36 | 88
  Bachelor's degree | 52 | 34 | 86
  Master's degree | 17 | 6 | 23
  Doctorate | 4 | 1 | 5
  Declined to answer | 1 | 0 | 1
Annual household income [Count of Participants; unit: Participants]
  Under $10,000 | 20 | 8 | 28
  $10,000 - $19,999 | 35 | 15 | 50
  $20,000 - $29,999 | 40 | 23 | 63
  $30,000 - $39,999 | 19 | 12 | 31
  $40,000 - $49,999 | 25 | 10 | 35
  $50,000 - $59,999 | 30 | 14 | 44
  $60,000 - $69,999 | 8 | 12 | 20
  $70,000 - $79,999 | 19 | 10 | 29
  $80,000 - $89,999 | 15 | 6 | 21
  Over $90,000 | 28 | 16 | 44
  Decline to answer | 53 | 19 | 72

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cigarette Abstinence
Description: Based on 1-item that asked "In the past 7 days, have you smoked any cigarettes?". The variable is coded 1 if they the participants indicated they did not smoke any cigarettes otherwise coded 0. A value of 1 = abstinence and 0 = not abstinent.
Time Frame: 1-month and 3-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Support2Quit App - Cognitive Dissonance Based Smoking Cessation | Comparison App - Smoking Cessation Support without Cognitive Dissonance Activities
Number analyzed (Participants) | 292 | 145
Participants
  1-Month Follow-Up | 102 | 38
  3-Month Follow-Up | 112 | 54
Statistical Analysis 1: Comparison: Support2Quit App - Cognitive Dissonance Based Smoking Cessation vs Comparison App - Smoking Cessation Support without Cognitive Dissonance Activities; This is a cross sectional analysis at 1-month; Test type: Superiority; p = .036, Regression, Logistic; Odds Ratio (OR) = 1.66, 95% CI 2-sided [1.04 to 2.67] — The Support2Quit group was scored 1 and the Comparison group was scored 0 (reference group for the odds ratio)
Statistical Analysis 2: Comparison: Support2Quit App - Cognitive Dissonance Based Smoking Cessation vs Comparison App - Smoking Cessation Support without Cognitive Dissonance Activities; This is a cross sectional analysis at 3-months; Test type: Superiority; p = .632, Regression, Logistic; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.72 to 1.72] — The Support2Quit group was scored 1 and the Comparison group was scored 0 (reference group for the odds ratio)

2. Primary Outcome: Fagerstrom Tobacco Dependence Scale
Description: This is a 6 item measure of tobacco dependence and response options are a mix of ordered categorical and dichotomous items. Item 1 "How many cigarettes per day to you smoke?" (0 = less than 10 cigarettes a day, 3 = 31 or more cigarettes a day). Item 2 "How soon after you wake do you smoke your first cigarette (0 = after 60 minutes, 3 = within 5 minutes). Item 3 "Is it hard to keep from smoking in places where it is prohibited (1 = yes, 0 = no). Item 4 "Which cigarette would you hate to give up most (1 = the first in the morning, 0 = any other). Item 5 "Do you smoke more cigarettes during the first 2 hours of the day compared to the rest of the day (1 = yes, 0 = no). Item 6 "Do you smoke when you are so ill you are in bed?" (1 = yes, 0 = no). A total sum score is computed and can range from 0 to 10 points with higher scores indicating higher levels of tobacco dependence.
Time Frame: Baseline, 1-month follow-up, 3-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Support2Quit App - Cognitive Dissonance Based Smoking Cessation | Comparison App - Smoking Cessation Support without Cognitive Dissonance Activities
Number analyzed (Participants) | 292 | 145
units on a scale
  Baseline | 5.7 (2.0) | 5.4 (1.9)
  1-Month Follow-Up | 4.1 (2.4) | 4.4 (2.2)
  3-Month Follow-Up | 4.0 (2.1) | 4.2 (2.4)
Statistical Analysis 1: Comparison: Support2Quit App - Cognitive Dissonance Based Smoking Cessation vs Comparison App - Smoking Cessation Support without Cognitive Dissonance Activities; This is a longitudinal analysis from baseline to 3-month follow-up; Test type: Superiority; p = .437, t-test, 2 sided; Mean Difference (Final Values) = -0.06, Standard Error of Mean 0.08 — The Support2Quit group was scored 1 and the Comparison group was scored 0 (reference group for the condition by time interaction)

3. Primary Outcome: Number of Participants With Reduction in Number of Cigarettes Smoked Per Day
Description: Represents whether or not (1 = yes, 0 = no) a reduction of cigarettes smoked per day is reported from the baseline assessment. A higher score indicates a reduction in cigarettes smoked.
Time Frame: 1-month and 3-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Support2Quit App - Cognitive Dissonance Based Smoking Cessation | Comparison App - Smoking Cessation Support without Cognitive Dissonance Activities
Number analyzed (Participants) | 292 | 145
Participants
  1-Month Follow-Up | 191 | 91
  3-Month Follow-Up | 218 | 110
Statistical Analysis 1: Comparison: Support2Quit App - Cognitive Dissonance Based Smoking Cessation vs Comparison App - Smoking Cessation Support without Cognitive Dissonance Activities; This is a cross sectional analysis at 1-month; Test type: Superiority; p = .088, Regression, Logistic; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.94 to 2.42] — The Support2Quit group was scored 1 and the Comparison group was scored 0 (reference group for the odds ratio)
Statistical Analysis 2: Comparison: Support2Quit App - Cognitive Dissonance Based Smoking Cessation vs Comparison App - Smoking Cessation Support without Cognitive Dissonance Activities; This is a cross sectional analysis at 3-months; Test type: Superiority; p = .646, Regression, Logistic; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.64 to 2.07] — The Support2Quit group was scored 1 and the Comparison group was scored 0 (reference group for the odds ratio)

4. Primary Outcome: Number of Participants With Reduction in the Number of Cigarettes Smoked Per Day and Reduced to 0-5 Cigarettes
Description: Represents whether or not (1 = yes, 0 = no) a reduction of cigarettes smoked per day is reported from the baseline assessment and is the number of daily cigarettes in 0-5 per day. A higher score indicates a reduction in cigarettes smoked per day and the number smoked is 5 or less.
Time Frame: 1-month and 3-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Support2Quit App - Cognitive Dissonance Based Smoking Cessation | Comparison App - Smoking Cessation Support without Cognitive Dissonance Activities
Number analyzed (Participants) | 292 | 145
Participants
  1-Month Follow-Up | 144 | 56
  3-Month Follow-Up | 165 | 74
Statistical Analysis 1: Comparison: Support2Quit App - Cognitive Dissonance Based Smoking Cessation vs Comparison App - Smoking Cessation Support without Cognitive Dissonance Activities; This is a cross sectional analysis at 1-month; Test type: Superiority; p = .010, Regression, Logistic; Odds Ratio (OR) = 1.77, 95% CI 2-sided [1.15 to 2.72] — The Support2Quit group was scored 1 and the Comparison group was scored 0 (reference group for the odds ratio)
Statistical Analysis 2: Comparison: Support2Quit App - Cognitive Dissonance Based Smoking Cessation vs Comparison App - Smoking Cessation Support without Cognitive Dissonance Activities; This is a cross sectional analysis at 3-months; Test type: Superiority; p = .158, Regression, Logistic; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.89 to 2.11] — The Support2Quit group was scored 1 and the Comparison group was scored 0 (reference group for the odds ratio)

ADVERSE EVENTS:
Time Frame: Data was collected from the baseline assessment to the 3 month post-baseline follow up assessment.
Description: Participants completed questionnaires at baseline, 1 month post-baseline and 3 months post-baseline.
Groups:
- Comparison App - Smoking Cessation App without Cognitive Dissonance Activities: This group will use an app that consists of tips for quitting cigarettes but does not include the cognitive dissonance component.
  Tips for Smoking Cessation App: App containing daily tips for smoking cessation
Arm/Group | Support2Quit App - Cognitive Dissonance Based Smoking Cessation | Comparison App - Smoking Cessation App without Cognitive Dissonance Activities
All-Cause Mortality (participants affected / at risk) | 0/292 | 0/145
Serious Adverse Events (participants affected / at risk) | 0/292 | 0/145
Other Adverse Events (participants affected / at risk) | 0/292 | 0/145

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-08-09): https://cdn.clinicaltrials.gov/large-docs/55/NCT05797155/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT05797155/SAP_001.pdf
  • Informed Consent Form (2024-03-06): https://cdn.clinicaltrials.gov/large-docs/55/NCT05797155/ICF_002.pdf